CLINICAL TRIAL: NCT03162718
Title: A Feasibility Study of Unsupervised, Pre-operative Exercise Program for Patients Scheduled for Lung Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Norris Cotton Cancer Center (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, Scientist, Psychiatry Research, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D17044
Record Dates: First submitted 2017-05-04; First posted 2017-05-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; exercise; pre-operative exercise program
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The investigators propose a mixed methods,16 single arm feasibility study of an unsupervised, pre-operative exercise prescription (uPEP) augmented by a wearable fitness device. The proposed study of 30 patients scheduled for lung cancer surgery will identify the strengths, weaknesses, and utility of this approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — single arm feasibility study of an unsupervised, pre-operative exercise prescription (uPEP) augmented by a wearable fitness device.

SUMMARY:
The paradigm of pre-operative exercise as a neoadjuvant therapy to reduce morbidity is increasingly promoted within general surgery and surgical oncology.

Patients with lung cancer participating in pre-operative exercise have better aerobic capacity and pulmonary function and shorter hospital length-of-stay after surgery. Additionally, pre-operative exercise may increase the likelihood of resuming exercise post-surgery, thereby accelerating the pace of rehabilitation and recovery.

In order to translate the research findings into sustainable clinical practice, clinician-scientists need to develop pragmatic and effective home-based exercise protocols. Wearable fitness devices offer a way to approximate the supervision that occurs in exercise research.

Before the investigators can develop an intervention in which patients receive tailored support similar to what occurs with supervised exercise, they need to pilot test the monitoring aspect of the wearable fitness device in conjunction with the pre-operative exercise program. The investigators propose a mixed methods, 16 single arm feasibility study of an unsupervised, pre-operative exercise prescription (uPEP) augmented by a wearable fitness device. The proposed study of 30 patients scheduled for lung cancer surgery will identify the strengths, weaknesses, and utility of this approach.

DETAILED DESCRIPTION:
The investigators propose a parallel mixed methods, 16 single arm, pre-post study with 30 participants scheduled for lung cancer surgery. At time of enrollment (at least 3 weeks before their scheduled surgery), participants will complete baseline assessments, receive the uPEP exercise prescription, and be oriented to the wearable fitness device. A research assistant will call the participant to conduct an audiotaped semi-structured interview regarding the acceptability of the electronically-monitored uPEP within 7- 14 days of enrollment. The study team will complete follow-up assessments on the day of surgery, two weeks after surgery, and four months after surgery. Data will also be collected from chart review and the wearable fitness device throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* This study will recruit English-speaking patients who:

  1. Are over the age of 18 and diagnosed with Stage I-III lung cancer;
  2. Are able to tolerate surgery (i.e., segmentectomy, lobectomy or bilobectomy) as indicated by standard clinical pre-op evaluation, including pulmonary function tests and cardiac evaluation (if indicated);
  3. Access to either Wi-Fi or cellular service and permission/ability to download the wearable fitness device app on an apple device, android, or computer (or willingness to use a study-provided iPod to allow the data to be uploaded to the study team);
  4. Are able to provide voluntary, written consent.

Exclusion Criteria:

* Participants will be excluded based on electronic health record (EHR) review (after obtaining HIPAA waiver) if they:

  1. Have a life expectancy of < 12 months or are receiving hospice services;
  2. Have a psychiatric diagnosis that would require significant study modification to meet their needs such as uncontrolled severe mental illness, substance abuse, or active suicidal ideation;
  3. Exhibit American College of Sports Medicine contraindications to exercise which include a resting heart rate of >120bpm, blood pressure >180/100mmHg or unstable angina;31
  4. Are unable to walk or to complete the 6-minute walk test. According to our current standard of care, those participants will be referred to physical therapy for evaluation and treatment and will be excluded from the study as unsupervised exercise would not be safe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Adherence to exercise: | Time 3, day of surgery
  number of completed pre-operative exercise sessions divided by number of prescribed sessions, according to exercise log

SECONDARY OUTCOMES:
Feasibility of recruitment: | Time 5, 16 weeks post-surgery
  number of patients enrolled divided by number of patients eligible
Acceptance of technology | Time 3, day of surgery
  number of hours the fitness tracker was worn in pre-operative period
Participant perception of exercise program | Time 2, 3-5 days before surgery
  semi-structured interview regarding perceptions of the exercise program
Participant perception of fitness tracker | Time 2, 3-5 days before surgery
  semi-structured interview regarding perceptions of the fitness tracker
Subjective minutes spent in exercise | Time 3, day of surgery
  Number of minutes spent in exercise according to exercise log
Objective minutes spent in exercise: | Time 3, day of surgery
  Number of minutes spent in exercise according to fitness tracker
Aerobic capacity: | Time 3, day of surgery
  Six minute walk test
Pulmonary function: | Time 2, 3-5 days before surgery
  Diffusion of lungs for carbon monoxide test
Subjective physical function: | Time 2, 3-5 days before surgery
  PROMIS (Patient-Reported Outcomes Measurement Information System) physical function scale
Objective physical function: | Time 3, day of surgery
  Grip strength per dynamometer
Length of stay in hospital: | Time 4, 2 weeks post-surgery
  Number of days from surgery to discharge home
Feasibility of Retention | 16 weeks post-surgery
  Number of patients completing all study assessments divided by the number enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen D Lyons, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center; David J Finley, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Finley DJ, Stevens CJ, Emond JA, Batsis JA, Fay KA, Darabos C, Sacks OA, Cook SB, Lyons KD. Potential effectiveness of a surgeon-delivered exercise prescription and an activity tracker on pre-operative exercise adherence and aerobic capacity of lung cancer patients. Surg Oncol. 2021 Jun;37:101525. doi: 10.1016/j.suronc.2021.101525. Epub 2021 Mar 5. PMID 33813267
- [Derived] Finley DJ, Fay KA, Batsis JA, Stevens CJ, Sacks OA, Darabos C, Cook SB, Lyons KD. A feasibility study of an unsupervised, pre-operative exercise program for adults with lung cancer. Eur J Cancer Care (Engl). 2020 Jul;29(4):e13254. doi: 10.1111/ecc.13254. Epub 2020 May 29. PMID 32469129